CLINICAL TRIAL: NCT02926248
Title: Effect of Colchicine on Range of Motion After Manipulation Under Anesthesia for the Stiff Total Knee Replacement: A Prospective Randomized Controlled Trial
Brief Title: Effect of Colchicine on Range of Motion After Manipulation Under Anesthesia for the Stiff Total Knee Replacement
Acronym: Colchine MUA
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Continuing IRB review was not submitted. Study was inactivated with the institutional IRB.
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-707
Record Dates: First submitted 2016-06-24; First posted 2016-10-06 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Manipulation Under Anesthesia
Keywords: Arthrofibrosis
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine (Experimental): Manipulation under Anesthesia (MUA) will be performed prior to 12 weeks after the index TKA. Patients will be randomized to oral colchicine 0.6 mg twice daily for 6 weeks. All patients will follow a standardized post-MUA physical therapy protocol.
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Manipulation under Anesthesia (MUA) will be performed prior to 12 weeks after the index TKA. Patients will be randomized to oral placebo twice daily for 6 weeks. All patients will follow a standardized post-MUA physical therapy protocol.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine is an anti-fibrotic and anti-inflammatory drug
  Other Names: Colcrys
  Arms: Colchicine
Other: Placebo
  Arms: Placebo

SUMMARY:
The specific aim of this study is to evaluate the effect of oral colchicine in primary TKA patients at 3 months following a manipulation under anesthesia.

DETAILED DESCRIPTION:
Adult primary unilateral TKA patients with less than 90° of knee flexion between 5 and 12 weeks after their index surgery will be screened for trial eligibility based on the inclusion and exclusion criteria above. Only patients from the protocol surgeons will be eligible to participate in this trial. MUA will be performed prior to 12 weeks after the index TKA. Patients will be randomized to either oral colchicine 0.6 mg twice daily for 6 weeks (treatment arm) or to oral placebo twice daily for 6 weeks in the placebo arm. All patients will follow a standardized post-MUA physical therapy protocol. Data will be collected prospectively, including study data collection sheets and medication diary. Other data sources will include office and inpatient medical records, operative reports, physical therapy records, hospital picture archiving and communication system (PACS) and radiology records. Outcomes will be collected at MUA, 6 weeks, 3 months, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral TKA indicated for MUA (knee flexion angle less than 90°)
* Primary Diagnosis of OA for TKA
* MUA indicated within 5 to 12 weeks of primary surgery
* Age greater than or equal to 18 years
* Patients with less than 10 degrees of a flexion contracture

Exclusion Criteria:

* Patients who are wheelchair bound
* Patients requiring concomitant arthroscopic or open procedures
* Revision TKA
* Patients requiring bilateral MUA
* Patients with renal disease (Creatinine > 1.5, and/or estimated creatinine clearance less than 30 mL/min)
* Patients with hepatic disease (known liver disease, cirrhosis, and/or AST/ALT>60)
* Patients concurrently taking strong CYP3A4 inhibitors:

  * Atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, amprenavir, aprepitant, diltiazem, erythromycin, fluconazole, fosamprenavir, grapefruit juice, verapamil
* Patients concurrently taking strong P-glycoprotein inhibitors:

  * Cyclosporine, ranolazine
* Patients concurrently taking medications that increase the risk for myopathy and rhabdomyolysis:

  * atorvastatin, fluvastatin, pravastatin, simvastatin, fibrates, gemfibrozil, digoxin
* Patients with a history of blood dyscrasias
* Pregnant patients
* Patients who are nursing mothers
* Patients with reported allergy to colchicine
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-03-21 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in Range of Motion | Change from baseline to 3 months post-operative
  Measured in Degrees by a goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No